CLINICAL TRIAL: NCT02687659
Title: TEMIS: a Pilot Study to Evaluate a Device to Characterize Ambulatory Physical Activity
Acronym: TEMIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Collaborators: University Hospital, Toulouse (Other); MEDES Institut de Médecine et de Physiologie Spatiales, Toulouse (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2014-A00444-43
Record Dates: First submitted 2014-05-31; First posted 2016-02-22 (Estimated); Last update posted 2016-02-22 (Estimated); Status verified 2016-02

CONDITIONS: Healthy; Sedentary
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Study group using TEMIS system (Experimental): using TEMIS system during physical exercises: walking, biking, running
  Interventions: Device: TEMIS system

INTERVENTIONS:
Device: TEMIS system — Wearing TEMIS system over the day during one week

SUMMARY:
Physical inactivity is a major public health issue. Prescription of physical activity appears necessary in some situation with cardiovascular risk. It is important to both qualify and quantify daily physical activity.

The aim of this project is to evaluate the TEMIS system (based on a smart T-shirt) performance in 12 healthy subjects, wearing this system over the daytime during one week.

DETAILED DESCRIPTION:
Healthy subjects have to make different physical activities, wearing the TEMIS system like slow and fast walking, biking, running.

ELIGIBILITY:
Inclusion Criteria:

* Men or women 18 - 50 yo
* BMI between 18 and 30
* Without chronic disease or chronic treatment (oral contraception is allowed)
* Normal electrocardiogram
* Able to do all the specified physical activity requested by the protocol
* Able to use smart phone and computers
* With access to WIFI, bicycle, and car
* Living in the close area
* Affiliated to public health insurance

Exclusion Criteria:

* Severe allergia
* Severe skin lesions at the thorax level
* Not able to use correctly the TEMIS system
* Will take plane during the week of evaluation
* Under protection

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2014-05; Primary Completion 2014-12 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
concordance (kappa score) between actual and estimated physical activity | One week (average of each day recording)
  Investigators will during the seven days of the protocol, when the system TEMIS is hold, evaluate the concordance between the activity really performed by the subject (questionnaire) and the activity calculated by the TEMIS System (Kappa test). Investigators will evaluate the following activity:
  lying position, sitting position, standing position, walking activity, running activity, bicycle activity, use of a vehicle (car, bus)

SECONDARY OUTCOMES:
total duration of recording in hours | One week (sum of each day recording)
number of subjects with adverse events | one week
  will be considered as adverse events
  * allergia
  * discomfort with removal of the system

CONTACTS AND LOCATIONS:
Overall Officials: Marc-Antoine CUSTAUD, MD, PhD, Principal Investigator — University Hospital, Angers
Locations (1):
- CHU Angers, Angers, Maine et Loire, France